CLINICAL TRIAL: NCT00724685
Title: Interest of Continuous Ropivacaine Administration Through an Elastomeric Pump (Pain Buster ) for the Surgery of Latissimus Dorsi and Serratus Micro Anastomotic Flaps
Brief Title: Interest of Continuous Ropivacaine Administration Through an Elastomeric Pump (Pain Buster) for the Surgery of Latissimus Dorsi and Serratus Micro Anastomotic Flaps
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRD07/3-Y; Eudract 2007-002983-89
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Post Operative Analgesia
Keywords: Ropivacaine; elastomeric pump; patient controlled analgesia; morphine consumption
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Active (Experimental)
  Interventions: Drug: Naropeine (Ropivacaine)

INTERVENTIONS:
Drug: Naropeine (Ropivacaine)
  Arms: Active
Drug: Placebo — saline
  Arms: Placebo

SUMMARY:
Continuous bupivacaine administration through an elastomeric pump (Pain Buster) has been found effective for post operative analgesia in a large range of surgery. Ropivacaine is a less toxic drug, never tested in the surgery of latissimus dorsi and serratus micro anastomotic flaps (from the investigators knowledge). The aim of the study is to evaluate the usefulness of this drug and device for post operative analgesia, associated with patient controlled analgesia with morphine. For this purpose a controlled randomized double blind trial against placebo (saline) is performed, enrolling 40 (20x2) patients during 3 years, in order to measure total morphine consumption during the first 48 post operative hours and to evaluate analgesia and sides effects of morphine in each group.

ELIGIBILITY:
Inclusion Criteria:

* operated for latissimus dorsi and serratus micro anastomotic flaps.
* 18 to 75 years old
* ASA I-II
* hospitalized in Nantes CHU Burns ICU
* giving their written informed consent
* with healthcare protection

Exclusion Criteria:

* declining the study
* with known sides effects with morphine and local anesthetics
* with known allergy or other reaction with used drugs
* with disease incompatible with anaesthetic procedure
* under law protection
* taking antiepileptic or antidepressant drugs
* pregnant (not any gender criteria)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | H 48

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Nantes, France